CLINICAL TRIAL: NCT00004176
Title: A Phase II Evaluation of Ethyol as an Esophageal Mucosal Protectant in the Treatment of Limited Disease Small Cell Lung Cancer With Chemotherapy and Twice-Daily Radiation
Brief Title: Amifostine, Chemotherapy, and Radiation Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067202; WU-98-0206; ALZA-WU-98-0206; NCI-V99-1559
Record Dates: First submitted 2000-01-21; First posted 2004-05-25 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Lung Cancer; Radiation Toxicity
Keywords: limited stage small cell lung cancer; drug/agent toxicity by tissue/organ; radiation toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Radiation Injuries | interventions — Amifostine; Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as amifostine may protect normal cells from the side effects of chemotherapy and radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of amifostine plus chemotherapy and radiation therapy in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the incidence and duration of moderate and severe acute esophagitis in patients with limited stage small cell lung cancer treated with amifostine chemoprotection plus chemotherapy and radiotherapy. II. Determine the tumor response to this regimen in these patients.

OUTLINE: Course 1: Patients receive amifostine IV over 5 minutes daily, followed by radiotherapy twice daily Monday through Friday for 3 weeks. Patients receive cisplatin IV over 30-60 minutes on day 1, and etoposide IV over 1 hour on days 1, 2, and 3. Courses 2-4: Patients receive amifostine over 15 minutes on day 1, followed by cisplatin IV over 30-60 minutes and etoposide IV over 1 hour every 3 weeks. Patients are followed at 1 month, then every 3 months until death.

PROJECTED ACCRUAL: Approximately 33 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed limited stage small cell lung cancer confined to one hemithorax Measurable disease No pleural effusion(s)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 75,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT and alkaline phosphatase no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Calcium normal (8.9-10.3 mg/dL) Cardiovascular: No history of congestive heart failure or myocardial infarction within the past 6 months No uncontrolled or unexplained rhythm disturbance or symptoms of unstable ischemic heart disease Other: Not pregnant Fertile patients must use effective contraception No prior or concurrent malignancy within the past 5 years, except: Basal or squamous cell skin cancer Carcinoma in situ of the cervix No concurrent infection No significant uncontrolled hyponatremia No other significant concurrent medical or psychiatric illness which would preclude compliance No antecedent hearing loss Afebrile for at least 3 days unless fever due to tumor or obstructive pneumonia

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified Other: No drugs that could potentiate nephrotoxicity of cisplatin (e.g., aminoglycosides or lithium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 1998-10; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H. Read, M.D., Study Chair — Washington University School of Medicine
Locations (4):
- United States (4):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania